CLINICAL TRIAL: NCT07152418
Title: A Study on the Therapeutic Efficacy of Monoclonal Antibody Drugs for Alzheimer's Disease Based on PET Research
Brief Title: Therapeutic Efficacy of Monoclonal Antibody Drugs for Alzheimer's Disease Based on PET Research
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0466
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease (AD); Alzheimer Dementia; Mild Cognitive Impairment (MCI)
Keywords: Alzheimer Disease; lecanemab; Tau PET; Aβ PET
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — lecanemab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lecanemab treatment group: Lecanemab 10 mg/kg
  Interventions: Biological: Lecanemab 10 mg/kg
- Conventional anti-dementia treatment: Early-stage Alzheimer's disease (AD) patients routinely take cholinesterase inhibitors such as donepezil for treatment.
  Interventions: Drug: Conventional anti-dementia treatment group

INTERVENTIONS:
Biological: Lecanemab 10 mg/kg — Lecanemab Injection Concentrate Solution (active ingredient at 100 mg/mL) is provided as a sterile aqueous solution containing 100 mg/mL of Lecanemab, 50 mmol/L citric acid, 350 mmol/L arginine/arginine hydrochloride, and 0.05% (w/v) polysorbate 80, with a pH of 5.0, and each vial is capable of being drawn into a volume of 5 mL. Lecanemab is to be administered via intravenous infusion over 60 minutes in saline solution. Lecanemab must be administered using an infusion system that includes a terminal 0.22 μM inline filter. The dosage of Lecanemab is 10 mg/kg.
  Groups: Lecanemab treatment group
Drug: Conventional anti-dementia treatment group — Conventional anti-dementia treatment: Early-stage Alzheimer's disease (AD) patients routinely take cholinesterase inhibitors such as donepezil for treatment.
  Groups: Conventional anti-dementia treatment

SUMMARY:
Preliminary clinical trial results indicate that Aβ-targeting monoclonal antibody drugs can delay disease progression more effectively. However, some patients still progress slowly to the moderate stage during treatment despite maintaining low Aβ/tau pathological protein loads. For such cases, patients and their families are fully informed about the potential lack of efficacy with continued treatment, and the decision is left to their discretion. Information regarding whether treatment is continued is documented and followed up to determine whether sustained benefits can be achieved. Previous further studies on lecanemab suggest that patients with low or absent tau pathology derive more significant clinical benefits, though large-sample validation remains lacking. This project will therefore enroll patients at clinical stages 3-4 (0.5 ≤ CDR ≤ 1) and monitor those progressing to moderate AD (CDR = 2) during monoclonal antibody therapy. Using tau pathology stratification, the study aims to identify which AD patients are most suitable for monoclonal antibody treatment and evaluate whether therapy continuation yields sustained benefits in patients progressing to moderate dementia, as well as whether patient selection should integrate both pathological (a-c stage) and clinical diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for Mild Cognitive Impairment (MCI) due to Alzheimer's Disease or mild-to-moderate AD. [Clinical Scores: CDR Global Score = 0.5 (for MCI) or 1 (for mild AD), corresponding to clinical stages 3-4, with a positive PIB-PET scan confirming amyloid pathology]
* Male or Female
* Between 50 and 85 years old (inclusive)
* Not currently participating in any other clinical trial or research study
* Participants must provide informed consent for this trial prior to enrollment and must voluntarily sign a written informed consent form
* Participants must be able to communicate effectively with the investigator and are expected to comply with the study requirements to completion

Exclusion Criteria:

* Any contraindication to MRI
* History of seizure within the past 6 months or refractory epilepsy.
* Unstable or severe psychiatric illness within the past 6 months.
* History of bleeding disorders, coagulopathy, or clinically significant coagulation abnormalities (e.g., platelet count <50,000/μL or INR >1.5).
* Uncontrolled diabetes mellitus or hypertension.
* History of unstable angina, myocardial infarction, advanced heart failure, or clinically significant conduction abnormalities within the past year.
* Active cancer treatment (e.g., chemotherapy, biologics, or radiation therapy), except maintenance therapy for cancers in remission (e.g., anti-estrogen therapy for breast cancer).
* Immunological disorders requiring ongoing immunosuppression, immunoglobulin therapy, monoclonal antibodies, or plasmapheresis.
* Breastfeeding individuals or women of childbearing potential not using highly effective contraception.
* History of severe allergic, anaphylactic reactions, or hypersensitivity to any inactive ingredients.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included early AD patients treated with Lecanemab and Conventional Anti-Dementia Treatment at the Second Affiliated Hospital of Zhejiang University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Aβ-PET centiloid values | Baseline, 18 months
  Statistical Comparison of Lecanemab versus Conventional Anti-Dementia Treatment Based on Aβ-PET Centiloid Scores

SECONDARY OUTCOMES:
Change from Baseline in the CDR at 18 Months | Baseline, 18 months
  Assessment of the Statistical Difference in CDR Scores Between Lecanemab and Conventional Anti-Dementia Treatment Groups
Change from Baseline in the MMSE at 18 Months | Baseline, 18 months
  Assessment of the Statistically Significant Difference in MMSE Scores Between Lecanemab and Conventional Anti-Dementia Treatment Groups
Change from Baseline in the MoCA at 18 Months | Baseline, 18 months
  Assessment of the Statistically Significant Difference in MoCA Scores Between Lecanemab and Conventional Anti-Dementia Treatment Groups
Change from Baseline in the NPI at 18 Months | Baseline, 18 months
  Assessment of the Statistically Significant Difference in NPI Scores Between Lecanemab and Conventional Anti-Dementia Treatment Groups
Blood AD molecular pathology | Baseline, 6 months, 12 months, 18 months
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using Plasma AD biomarkers (Aβ42, Aβ42/Aβ40, T-tau, P-tau181, P-tau231, P-tau217, NFL levels)

IPD SHARING:
Plan to Share IPD: Undecided